CLINICAL TRIAL: NCT02072655
Title: Impact of Socio-aesthetic Care in the Quality of Life of Patients Treated for Lymphoma During and After Hospitalization
Acronym: CareSSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AOI PM 2012-12
Record Dates: First submitted 2014-02-20; First posted 2014-02-26 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

ARMS (2):
- without socio-asthetic care (No Intervention)
- with socio-aesthetic cares (Experimental)
  Interventions: Procedure: socio-aesthetic care

INTERVENTIONS:
Procedure: socio-aesthetic care — * care of the face
  * skin cleansing with cleansing milk to remove impurities
  * a gentle scrub to exfoliate and cleanse the skin
  * a relaxing massage
  * moisturizing mask
  * application of a moisturizer suited to specific patient skin: skin reactivity, dehydration ...
  * care manicure / pedicure,
  * massages
  * makeup, advice (scarves, wigs care products adapted to the skin changes ...) and helping relationship.
  Arms: with socio-aesthetic cares

SUMMARY:
In the early 2000s , professional and patient organizations are mobilizing to highlight the psychosocial impact of cancer disease , not only during but also after the acute phase.

In 2003, the government launched the Cancer Plan I reinforced in December 2011 by the Cancer Plan II whose objectives include : " Develop a personalized care taking into account the pain and psychological and social support " and " increase opportunities for patients to benefit from supportive care "and" promote the professional integration .

This study aims to show that beyond the immediate benefits of the social aesthetic cares in hospital (direct soothing, improving the quality of the skin injured by chemotherapy , feeling of escape ... ), these treatments can also affect quality of life for patients during and after hospitalization. They also may have an impact on the maintenance of social and / or professional satisfactory throughout the planned chemotherapy aplastic period .

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* Hospitalized in the Hematology care unit in UH Angers
* Initial Hodgkin lymphoma, diffuse large B-cell lymphoma and mantle cell lymphoma
* Without previous socio-aesthetic care.

Exclusion Criteria:

* Age <18 years old.
* Patient protected by the law.
* Patient at end of life.
* Patient unable to respond to the questionnaire.
* Previous Socio aesthetic care.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Quality of life score | Change form baseline in Quality of life score at an average of 5 months (4 to 6 cycles of chemotherapy).
  * For patients in control group, arbitrarily during their fifth cycle of chemotherapy
  * For patients in interventional group during the course of chemotherapy after the third socio-aesthetic care, or at the latest, at the sixth treatment.

SECONDARY OUTCOMES:
Coopersmith Self-esteem inventory | Change form baseline in Coopersmith Self-esteem inventory score at an average of 5 months (4 to 6 cycles of chemotherapy).
Body Image Scale assessment | Change form baseline in body image scale assessment score at an average of 5 months (4 to 6 cycles of chemotherapy).
Social life assessment | Change form baseline in social life assessment score at an average of 5 months (4 to 6 cycles of chemotherapy).

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Care Unit - UH Angers, Angers, France